CLINICAL TRIAL: NCT03668808
Title: Comparison of Insulin Degludec With Insulin Glargine U100 for Adults With Type 1 Diabetes Travelling Across Multiple Time Zones. A Pilot Study.
Brief Title: Comparison of Insulin Degludec With Insulin Glargine U100 for Adults With Type 1 Diabetes Crossing Multiple Time Zones.
Acronym: SafrTravlT1D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ISS-001227; U1111-1210-7350 (Registry Identifier: Universal Trial Number - World Health Organization (WHO))
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Insulin Degludec; Insulin Glargine; Air Travel; Continuous Glucose Monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Intervention Model Description: Subjects will begin in Honolulu, HI (HNL), fly to Newark (EWR) where they will stay for up to 72 hours followed by a return long-haul flight back to Honolulu with up to 72 hours at this destination. This journey will be repeated after a 2 week period when subjects return to their original insulin treatment regimen and then switch to the alternative basal insulin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Insulin Degludec (Experimental): Subjects with type 1 diabetes and on multiple daily injections will use basal insulin Degludec and the TRESIBA® FLEXTOUCH® pens during a long-haul flight and randomized to this arm first or second.
  Interventions: Drug: Insulin Degludec; Device: TRESIBA® FLEXTOUCH®
- Insulin Glargine U100 (Active Comparator): Subjects with type 1 diabetes and on multiple daily injections will use basal insulin Glargine U100 and the LANTUS® SOLOSTAR® INSULIN PEN during a long-haul flight and randomized to this arm first or second.
  Interventions: Drug: Insulin Glargine; Device: LANTUS® SOLOSTAR® INSULIN PEN

INTERVENTIONS:
Drug: Insulin Degludec — Subjects will use Insulin Degludec (Tresiba) with TRESIBA® FLEXTOUCH® pens as their basal insulin during a 9-10 hour flight, at each destination, and then during a return flight.
  Other Names: Tresiba
  Arms: Insulin Degludec
Drug: Insulin Glargine — Subjects will use Insulin Glargine (Lantus) with LANTUS® SOLOSTAR® INSULIN PEN as their basal insulin during a 9-10 hour flight, at each destination, and then during a return flight.
  Other Names: Lantus
  Arms: Insulin Glargine U100
Device: TRESIBA® FLEXTOUCH® — Subjects will use Tresiba FlexTouch pens when using Tresiba as their basal insulin during a 9-10 hour flight, at each destination, and then during a return flight.
  Other Names: Insulin Degludec
  Arms: Insulin Degludec
Device: LANTUS® SOLOSTAR® INSULIN PEN — Subjects will use Lantus SoloStar insulin pens when using Lantus as their basal insulin during a 9-10 hour flight, at each destination, and then during a return flight.
  Other Names: Insulin Glargine
  Arms: Insulin Glargine U100

SUMMARY:
The purpose of the proposed study is to compare insulin Degludec [TRESIBA® (insulin degludec injection)] with insulin Glargine U100 [Lantus® (insulin glargine injection)] to determine the basal insulin of choice for adults with type 1 diabetes (T1D) who fly non-stop across multiple time zones. With the introduction of Degludec as basal insulin for T1D and the opportunity to vary time of injection between 8 and 40 hours, the use of Degludec as a basal insulin may make it easier for both people living with T1D and diabetologists to plan long-haul travel compared to the use of existing basal insulins when crossing multiple time zones.The study hypothesis is that once daily Degludec as the basal insulin will provide better glycemic control for people with type 1 diabetes on multiple daily injections who are traveling non-stop across multiple time zones than once daily Glargine U100.

DETAILED DESCRIPTION:
This study will be an open-label, single center, pilot study. Participants will be randomized to either Glargine U100 or Degludec as the basal insulin, then a 2 week break, and followed by a cross-over to the other insulin. Each study period will begin in Honolulu, Hawaii (HI) (airport code HNL) with a non-stop flight to Newark, New Jersey (NJ) (EWR) lasting approximately 10 hours with a 6 hour time difference between destinations. After up to 72 hours in EWR, participants will return to Honolulu and spend up to 72 hours at that destination. Investigators plan to recruit 25 adults with established T1D currently being treated with multiple daily injections of insulin (MDI).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥18 and ≤65 years of age.
2. Type 1 diabetes mellitus (diagnosed clinically and treated with multiple daily injections of insulin) for ≥12 months.
3. HbA1c <10% within 30 days of being enrolled in the study
4. Current treatment with any basal insulin analogue as the once daily basal insulin given in the evening (22) and no fewer than three injections with rapid acting bolus insulin (e.g. insulin aspart, insulin lispro, or insulin glulisine) as mealtime bolus insulin therapy.
5. No contraindication to long-haul travel.
6. No recurrent severe hypoglycemia (more than 1 severe hypoglycemic event requiring hospitalization during the last 12 months), or hypoglycemia unawareness as judged by a score of >4 on the Gold score (23), or hospitalization for diabetic ketoacidosis during the previous 6 months.
7. Willing and able to use a continuous glucose monitoring device (e.g. Dexcom G4).
8. Ability to self-manage insulin therapy (verbal confirmation at screening visit) of a changed bolus insulin dose the preceding 2 months prior to screening.
9. Ability and willingness to adhere to the protocol, including performance of self-monitored blood glucose (SMBG) readings and self-adjustment of insulin doses according to protocol.

   -

Exclusion Criteria:

1. Current use of an insulin pump.
2. Use within the last 3 months prior to enrollment visit 1 of any glucose-lowering drug other than insulin.
3. Initiation or significant change of any systemic treatment which, in the investigator's opinion, could interfere with glucose metabolism, such as systemic corticosteroids, beta-blockers or monoamine oxidase inhibitors (inhaled corticosteroids allowed).
4. Proliferative retinopathy or maculopathy requiring treatment, according to the investigator.
5. Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures.
6. Any clinically significant disease or disorder, which in the investigator's opinion could interfere with the results of the trial.
7. Mental incapacity, psychiatric disorder, unwillingness or language barriers precluding adequate understanding or cooperation, including subjects not able to read or write, and known or suspected abuse of alcohol, narcotics, or illicit drugs.
8. Known or suspected allergy to any of the trial products or related products.
9. Receipt of any investigational drug or participation in other trials within 1 month prior to Visit 1.

   -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2020-09-19 (Actual); Study Completion 2020-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kerr, M.D., Principal Investigator — Sansum Diabetes Research Institute
Locations (2):
- United States (2):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - inControl Diabetes Center, Honolulu, Hawaii

IPD SHARING:
Plan to Share IPD: Undecided
Undecided to whether to make individual participant data available.

REFERENCES:
- [Derived] Bevier WC, Castorino KN, Axelrod C, Haroush G, Farfan CC, Shelton N, Nelson K, Spink LA, Liu H, Kerr D. Traveling Across Time Zones With Type 1 Diabetes: A Pilot Study Comparing Insulin Degludec With Insulin Glargine U100. Diabetes Care. 2022 Jan 1;45(1):67-73. doi: 10.2337/dc21-1524. PMID 34716211

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 2018-2019, 25 subjects from the local community were screened for eligibility and then randomly assigned to one arm of the study . When the first arm was completed, the subjects crossed over to the other arm of the study.
Pre-assignment Details: 25 Participants were randomly assigned to one arm and then crossed over to the other arm when the first assignment was completed.
Groups:
- Insulin Degludec, Then Insulin Glargine: Subjects with type 1 diabetes and on multiple daily injections will use basal insulin Degludec and the TRESIBA® FLEXTOUCH® pens during a long-haul flight and randomized to this arm first or second.
  Insulin Degludec: Subjects will use Insulin Degludec (Tresiba) with TRESIBA® FLEXTOUCH® pens as their basal insulin during a 9-10 hour flight, at each destination, and then during a return flight.
  After a washout period of 2 weeks, the subjects crossed over to the other basal insulin, Insulin Glargine.
- Insulin Glargine U100, Then Insulin Degludec: Subjects with type 1 diabetes and on multiple daily injections will use basal insulin Glargine U100 and the LANTUS® SOLOSTAR® INSULIN PEN during a long-haul flight and randomized to this arm first or second.
  Insulin Glargine: Subjects will use Insulin Glargine (Lantus) with LANTUS® SOLOSTAR® INSULIN PEN as their basal insulin during a 9-10 hour flight, at each destination, and then during a return flight.
  After a washout period of 2 weeks, subjects crossed over to the other basal insulin, Insulin Degludec.
Period: First Intervention
Arm/Group | Insulin Degludec, Then Insulin Glargine | Insulin Glargine U100, Then Insulin Degludec
Started | 13 | 12
Completed | 11 | 10
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2
Period: Washout Period
Arm/Group | Insulin Degludec, Then Insulin Glargine | Insulin Glargine U100, Then Insulin Degludec
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Insulin Degludec, Then Insulin Glargine | Insulin Glargine U100, Then Insulin Degludec
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects randomly assigned to one arm and then crossed over to the other arm when the first was completed.
Groups:
- All Study Participants: Subjects with type 1 diabetes and on multiple daily injections will use either basal insulin Glargine U100 and the LANTUS® SOLOSTAR® INSULIN PEN or they will use basal insulin Degludec and the TRESIBA® FLEXTOUCH® pens during a long-haul flight and randomized to these arms first or second.
  For Insulin Glargine: Subjects will use Insulin Glargine (Lantus) with LANTUS® SOLOSTAR® INSULIN PEN as their basal insulin during a 9-10 hour flight, at each destination, and then during a return flight. After a washout period of 2 weeks, subjects crossed over to the other basal insulin, Insulin Degludec.
  For Insulin Degludec: Subjects will use Insulin Degludec (Tresiba) with TRESIBA® FLEXTOUCH® pens as their basal insulin during a 9-10 hour flight, at each destination, and then during a return flight. After a washout period of 2 weeks, the subjects crossed over to the other basal insulin, Insulin Glargine.
Arm/Group | All Study Participants
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Hypoglycemia awareness [Mean (Standard Deviation); unit: units on a scale] — Hypoglycemia awareness - ability to perceive onset of hypoglycemia in patients who use insulin to treat diabetes.
  "Gold Score" poses the question: "Do you know when your hypos are commencing?". Patients complete a 7 point Likert scale from 1 "always aware" to 7 "never aware." "Fear of Hypoglycemia scale" - a 33 question survey describing behaviors and worry about hypoglycemia. Questions are answered with 0 never, 1 rarely, 2 sometimes, 3 often, 4 almost always. Total range is 0 minimum to 132 maximum. Total scores (>50) indicate more fear of hypoglycemia.
  units on a scale
    Gold score | 2.0 (1.2)
    Fear of hypoglycemia scale | 36.6 (18.1)

OUTCOME MEASURES:

1. Primary Outcome: Continuous Glucose Monitoring - Time in Range (70-140 mg/dl)
Description: Time in range (70-140 mg/dl) [percentage of glucose readings or hours per day] by continuous glucose monitoring (CGM) during the initial 24 hours local time (starting within 2 hours after arriving) in Newark, NJ after flying 9-10 hours West to East (from Honolulu, HI) and after the return journey from Newark to Honolulu (flying East to West).
Time Frame: During the initial 24 hours local time and starting within 2 hours after arrival
Population: All participants (n=21) who completed both arms of the study were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of Time in Range 70-140mg/dL
Arm/Group | Insulin Degludec | Insulin Glargine U100
Number analyzed (Participants) | 21 | 21
percentage of Time in Range 70-140mg/dL
  Eastward travel | 36.3 (22.2) | 45.6 (21.1)
  Westward travel | 37.2 (22.2) | 43.9 (20.0)
Statistical Analysis 1: Comparison: Insulin Degludec vs Insulin Glargine U100; Null hypothesis is there was no difference in Time in Range (70-140mg/dl) in the initial 24 hours at destination, whether after Eastward travel or Westward travel, between Insulin Degludec & Insulin Glargine U100. Travel direction not tested. Criterion for significance set at 0.05; using paired t-test analysis, a sample size of 21 subjects would achieve a power of at least 77% to detect a difference of 10% between basal insulins assuming the standard deviation of the difference is <106 minutes; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was p=0.05

2. Secondary Outcome: Continuous Glucose Monitoring - Time in Range (70-180 mg/dl)
Description: Time in range (70-180 mg/dl) [percentage of glucose readings or hours per day] by continuous glucose monitoring (CGM) during the first 24 hours after arriving in HNL and EWR (starting within 2 hours after arrival).
Time Frame: During the initial 24 hours local time and starting within 2 hours after arrival
Measure: Mean (Standard Deviation); unit: percentage of Time in Range 70-180mg/dL
Arm/Group | Insulin Degludec | Insulin Glargine U100
Number analyzed (Participants) | 21 | 21
percentage of Time in Range 70-180mg/dL
  Eastward travel | 55.0 (21.7) | 62.3 (19.3)
  Westward travel | 54.5 (24.7) | 61.2 (24.7)
Statistical Analysis 1: Comparison: Insulin Degludec vs Insulin Glargine U100; Null hypothesis is there was no difference in Time in Range (70-180mg/dl) in the initial 24 hours at destination, whether after Eastward travel or Westward travel, between Insulin Degludec & Insulin Glargine U100. Travel direction not tested. Criterion for significance set at 0.05; using paired t-test analysis, a sample size of 21 subjects would achieve a power of at least 77% to detect a difference of 10% between basal insulins assuming the standard deviation of the difference is <106 minutes; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was p=0.05

3. Secondary Outcome: Mean ± SD CGM Glucose (mg/dl)
Description: Mean ± standard deviation of CGM glucose (mg/dl) by CGM during the flight and during the 72 hours at the destination
Time Frame: In flight period of time and for 72 hours at each destination
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Degludec | Insulin Glargine U100
Number analyzed (Participants) | 21 | 21
mg/dL
  In-flight eastward | 166.3 (55.2) | 158.8 (58.9)
  In-flight westward | 157.0 (37.5) | 146.1 (52.3)
  72 hours at destination after eastward travel | 154.3 (43.8) | 147.6 (34.0)
  72 hours at destination after westward travel | 160.4 (35.4) | 156.3 (34.6)
Statistical Analysis 1: Comparison: Insulin Degludec vs Insulin Glargine U100; Null hypothesis is there was no difference in Mean ± SD CGM glucose (mg/dl) in flight, East or West travel, and in 72 hours at destination, whether after East or West travel, between Insulin Degludec & Insulin Glargine U100. Travel direction not tested. Criterion for significance was at 0.05. Using paired t-test analysis, a sample size of 21 subjects would achieve a power of at least 77% to detect a difference of 10% between basal insulins assuming the SD of the difference is <106 minutes; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was p=0.05

4. Secondary Outcome: CGM % Time <70 mg/dl
Description: % time <70 mg/dl by CGM
Time Frame: In flight period of time and for 72 hours at each destination
Measure: Mean (Standard Deviation); unit: percentage of Time below range <70 mg/dL
Arm/Group | Insulin Degludec | Insulin Glargine U100
Number analyzed (Participants) | 21 | 21
percentage of Time below range <70 mg/dL
  Eastward travel in flight | 9.9 (21.5) | 8.9 (13.5)
  Westward travel in flight | 4.1 (7.3) | 9.9 (12.9)
  Eastward flight 72 hours at destination | 10.0 (9.6) | 10.5 (8.6)
  Westward flight 72 hours at destination | 8.4 (6.8) | 8.2 (6.9)
Statistical Analysis 1: Comparison: Insulin Degludec vs Insulin Glargine U100; Null hypothesis is that there was no difference in CGM % time <70 mg/dl in flight, East or West travel, and in 72 hours at destination, whether after East or West travel, between Insulin Degludec and Insulin Glargine U100. Travel direction not tested. Criterion for significance was at 0.05. Using paired t-test analysis, a sample size of 21 subjects would achieve a power of at least 77% to detect a difference of 10% between basal insulins assuming the SD of the difference is <106 minutes; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was p=0.05

5. Secondary Outcome: CGM % Time 70-180 mg/dl
Description: % time 70-180 mg/dl by CGM
Time Frame: In flight period of time and for 72 hours at each destination
Measure: Mean (Standard Deviation); unit: percentage of Time in Range 70-180mg/dL
Arm/Group | Insulin Degludec | Insulin Glargine U100
Number analyzed (Participants) | 21 | 21
percentage of Time in Range 70-180mg/dL
  Eastward travel in-flight | 50.5 (24.0) | 58.9 (30.8)
  Westward travel in-flight | 65.1 (23.6) | 64.0 (21.0)
  Eastward travel 72 hours at destination | 58.3 (18.8) | 62.0 (16.2)
  Westward travel 72 hours at destination | 56.7 (18.8) | 59.2 (23.0)
Statistical Analysis 1: Comparison: Insulin Degludec vs Insulin Glargine U100; Null hypothesis is that there was no difference in CGM % time 70-180 mg/dl in flight, East or West travel, and in 72 hours at destination, whether after East or West travel, between Insulin Degludec & Insulin Glargine U100. Travel direction not tested. Criterion for significance was at 0.05. Using paired t-test analysis, a sample size of 21 subjects would achieve a power of at least 77% to detect a difference of 10% between basal insulins assuming the SD of the difference is <106 minutes; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was p=0.05

6. Secondary Outcome: CGM % Time >180 mg/dl
Description: % time >180 mg/dl by CGM
Time Frame: In flight period of time and for 72 hours at each destination
Measure: Mean (Standard Deviation); unit: percentage of Time above Range >180mg/dL
Arm/Group | Insulin Degludec | Insulin Glargine U100
Number analyzed (Participants) | 21 | 21
percentage of Time above Range >180mg/dL
  In flight Eastward travel %Time above Range >180mg/dL | 39.5 (27.9) | 32.3 (31.5)
  In flight Westward travel %Time above Range >180mg/dL | 30.8 (25.4) | 26.0 (23.5)
  Eastward 72 hours at destination % Time above Range >180mg/dL | 31.7 (21.3) | 27.6 (17.2)
  Westward 72 hours at destination % Time above Range >180mg/dL | 34.9 (21.9) | 32.7 (23.1)
Statistical Analysis 1: Comparison: Insulin Degludec vs Insulin Glargine U100; Null hypothesis is that there was no difference in CGM % time >180 mg/dl in flight, East or West travel, and in 72 hours at destination, whether after East or West travel, between Insulin Degludec & Insulin Glargine U100. Travel direction not tested. Criterion for significance was at 0.05. Using paired t-test analysis, a sample size of 21 subjects would achieve a power of at least 77% to detect a difference of 10% between basal insulins assuming the SD of the difference is <106 minutes; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was p=0.05

7. Secondary Outcome: CGM - Coefficient of Variation (CV)
Description: Coefficient of variation of CGM values - glycemic variability (CV, %)
Time Frame: In flight period of time and for 72 hours at each destination
Measure: Mean (Standard Deviation); unit: percentage of Glycemic Variability %
Arm/Group | Insulin Degludec | Insulin Glargine U100
Number analyzed (Participants) | 21 | 21
percentage of Glycemic Variability %
  Eastward In-flight Glycemic variability CV % | 30.6 (15.9) | 31.0 (14.0)
  Westward In-flight Glycemic variability CV % | 28.2 (8.4) | 33.7 (10.1)
  Eastward 72-hours at destination Glycemic variability CV % | 39.9 (9.3) | 41.0 (10.8)
  Westward 72-hours at destination Glycemic variability CV % | 38.6 (7.4) | 39.5 (9.3)
Statistical Analysis 1: Comparison: Insulin Degludec vs Insulin Glargine U100; Null hypothesis is there was no difference in CGM - Coefficient of Variation (CV) in flight, East or West travel, and in 72 hours at destination, whether after East or West travel, between Insulin Degludec & Insulin Glargine U100. Travel direction not tested. Criterion for significance was at 0.05. Using paired t-test analysis, a sample size of 21 subjects would achieve a power of at least 77% to detect a difference of 10% between basal insulins assuming the SD of the difference is <106 minutes; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was p=0.05

8. Secondary Outcome: CGM Fasting Blood Glucose (FBG)
Description: Fasting Blood Glucose (FBG) was determined using CGM at each destination on the morning after arrival.
Time Frame: At 0600 local time on the morning after arrival at each destination
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Degludec | Insulin Glargine U100
Number analyzed (Participants) | 21 | 21
mg/dL
  After eastward travel | 143 (80) | 137 (60)
  After westward travel | 137 (60) | 140 (79)
Statistical Analysis 1: Comparison: Insulin Degludec vs Insulin Glargine U100; Null hypothesis is there was no difference in CGM Fasting Blood Glucose (FBG) at 0600 local time at destination, whether after East or West travel, between Insulin Degludec and Insulin Glargine U100. Travel direction not tested. Criterion for significance was set at 0.05, and using a paired t-test analysis, a sample size of 21 subjects would achieve a power of at least 77% to detect a difference of 10% between basal insulins assuming the standard deviation of the difference is <106 minutes; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was p=0.05

9. Secondary Outcome: Liverpool Jet-Lag Questionnaire
Description: This is a Questionnaire about jet-lag and fatigue administered at the destinations after arrival. Jet Lag is rated on a 0-10 scale (0 - insignificant jet lag to 10 - very bad jet lag). Fatigue is rated on a scale of -5 to +5 (more fatigue to less fatigue).
Time Frame: After 24 and 48 hours at the destination after arrival
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Insulin Degludec | Insulin Glargine U100
Number analyzed (Participants) | 21 | 21
score on a scale
  Eastward jet lag after 24 hours | 2.5 (2.6) | 4.1 (2.8)
  Eastward jet lag after 48 hours | 1.6 (2.7) | 3.8 (3.4)
  Eastward fatigue after 24 hours | 0.2 (1.6) | 0.2 (2.7)
  Eastward fatigue after 48 hours | -0.7 (1.8) | -1.5 (2.3)
  Westward jetlag after 24 hours | 3.2 (3.3) | 3.5 (3.3)
  Westward jetlag after 48 hours | 3.5 (2.9) | 2.9 (3.3)
  Westward fatigue after 24 hours | -1.6 (2.0) | -1.5 (2.3)
  Westward fatigue after 48 hours | 3.5 (2.9) | -0.7 (2.4)
Statistical Analysis 1: Comparison: Insulin Degludec vs Insulin Glargine U100; Null hypothesis is that there was no difference in Liverpool Jet-Lag Questionnaire after 24 and 48 hours at the destination, whether after Eastward travel or after Westward travel, between Insulin Degludec and Insulin Glargine U100. Travel direction not tested. The criterion for significance was set at 0.05, and using a paired t-test analysis, a sample size of 21 subjects would achieve a power of at least 77% to detect a difference of 10% between basal insulins; Test type: Superiority; p < 0.01, t-test, 2 sided — The threshold for statistical significance was p=0.05

10. Secondary Outcome: Sleep Quantity Measured by ActiGraph
Description: Measurement of sleep duration (TST - Total sleep time in minutes)
Time Frame: During 24 hours at each destination
Population: The pre-specified intent was to combine insulin arms if there were no differences between insulin arms. Sleep quantity was compared at each destination.
Measure: Median (Inter-Quartile Range); unit: Minutes
Groups:
- Sleep at Each Destination: Sleep quantity at each destination, either New York or Hawaii.
Arm/Group | Sleep at Each Destination
Number analyzed (Participants) | 21
Minutes
  Total sleep time, minutes in NY | 489 [390 to 572]
  Total sleep time, minutes in HI | 398 [337 to 422]
Statistical Analysis 1: Comparison: Sleep at Each Destination; Null hypothesis is that there was no difference in Sleep quantity measured by ActiGraph in 24 hours at the destination, whether after Eastward or after Westward travel, between Insulin Degludec and Insulin Glargine U100. Travel direction not tested. The criterion for significance was set at 0.05, and using a paired t-test analysis, a sample size of 21 subjects would achieve a power of at least 77% to detect a difference of 10% between basal insulins; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney) — The tests were performed with a significance level of 0.05 (two-sided)

11. Secondary Outcome: Sleep Efficiency Measured by ActiGraph
Description: Measurement of sleep efficiency (SE% - total sleep time in minutes divided by time in bed in minutes)
Time Frame: During 24 hours at each destination
Population: The pre-specified intent was to combine insulin arms if there were no differences between insulin arms. Sleep quality/efficiency was compared at each destination.
Measure: Median (Inter-Quartile Range); unit: percentage of total sleep/time in bed
Groups:
- Sleep at Each Destination: Sleep quality/efficiency at each destination, either New York or Hawaii.
Arm/Group | Sleep at Each Destination
Number analyzed (Participants) | 21
percentage of total sleep/time in bed
  SE% in NY | 92 [90 to 95]
  SE% in HI | 89 [86 to 94]
Statistical Analysis 1: Comparison: Sleep at Each Destination; Null hypothesis is there was no difference in Sleep efficiency measured by ActiGraph in 24 hours at the destination, whether after Eastward or after Westward travel, between Insulin Degludec and Insulin Glargine U100. Travel direction not tested. The criterion for significance was set at 0.05, and using a paired t-test analysis, a sample size of 21 subjects would achieve a power of at least 77% to detect a difference of 10% between basal insulins; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney) — The tests were performed with a significance level of 0.05 (two-sided)

ADVERSE EVENTS:
Time Frame: Up to 5 weeks for each intervention - basal insulin optimization and travel
Description: The study population included all participants who completed both arms of the study.
Arm/Group | Insulin Degludec, Then Insulin Glargine | Insulin Glargine U100, Then Insulin Degludec
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT03668808/Prot_SAP_000.pdf